CLINICAL TRIAL: NCT06894082
Title: COOPERATION BETWEEN THE MEDICAL ELECTRORADIOLOGY MANIPULATOR (MEM) AND THE RADIOLOGIST IN TUMOR IMAGING ASSESSMENTS: CIMER-IPC 2023-030
Brief Title: Study of Radiology Manipulator Work Validation by the Radiologist
Acronym: Cimer
Status: Recruiting | Type: Observational
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Other Study IDs: CIMER-IPC 2023-030; health data hub (Other: health data hub)
Record Dates: First submitted 2024-11-25; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Solid Cancer

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective of this study is to evaluate the pre-filling work on target and non-target lesions, and the detection of any new lesions reported by the MEM trained in protocol evaluations, in a structured table to prepare the radiologist's work in interpreting RECIST 1.1 scans.

To meet this objective, patients taking part in the CIMER study will first have been included in a research protocol requiring scans with RECIST 1.1 interpretation.

The Baseline examination will be performed and interpreted according to RECIST 1.1 without informing the radiologist performing the reading that the patient is included in the study, so as not to introduce an interpretation bias.

During the first evaluation. The investigating MEM alone will carry out a preliminary analysis of the first evaluation and will present his results to the radiologist in charge of the evaluation, who will validate the conformity of the results.

DETAILED DESCRIPTION:
In recent years, imaging has become essential in the evaluation of treatment efficacy in medical oncology . As a result, the proportion of clinical trials involving imaging has risen sharply, and radiology departments are faced with the problem of work overload in the face of complex specific interpretation methods which have developed further recently with immunotherapies (iRECIST 2017, imRECIST 2018).

The RECIST 1.1 method is the reference method for evaluating treatments of solid cancers because it allows standardization, reproducibility and a common language between all stakeholders.

Interpretation is based on :A pre-treatment examination called Baseline, which defines the lesions to be monitored and evaluation examinations (generally every 6 weeks) to compare measurements and define overall tumor evolution (Complete Response, Partial Response, Stable Disease, Progressive Disease).

It is difficult to concentrate the increasing number of protocol examinations on a small number of radiologists. As a result, the number of radiologists involved in these assessments multiplies the difficulties and risks of error. For the past 2 years, the Institut Paoli Calmettes has been testing cooperative protocol readings between radiologists and medical electroradiology manipulators (MEMs). First impressions are encouraging, and show that both radiologists and investigators are satisfied, with a priori an increase in the quality of radiological reports and a saving in interpretation time that we hope to objectify. This type of organization has already been partly studied in other Cancer Centers, such as the Centre Antoine Lacassagne in Nice and the Centre Henri Becquerel in Rouen, demonstrating the effectiveness of manipulators in measuring target lesions.

Artificial Intelligence solutions are currently being developed in all areas of imaging, opening up the possibility of applications to RECIST assessments). While these solutions appear to be of interest for the reassessment of previously identified lesions, their limitations for the time being relate to the differentiation between malignant lesions and benign tissue. The aim of adding AI to human analyses would be to further improve measurement performance and speed of assessment, without replacing but implementing the contribution that specialized manipulators could already make to radiological interpretations. In a difficult period for the radiology manipulator profession, these proposed new skills may also give new interest to the profession by integrating into an advanced practice pathway for which radiologists remain responsible. The aim of this study is to evaluate the contribution of collaboration with a manipulator specialized in therapeutic trials for the radiologist in charge of interpretation.

It aims to redefine the sharing of activities between delegators (mainly doctors) and other healthcare professionals (receiving delegation, or delegates), by entrusting the latter with certain activities outside their usual remit, in order to free up medical time while making the careers of these healthcare professionals more attractive.

The innovative nature of this cooperation would highlight the value of radiologist/EMM collaboration in intellectual acts.

It is not possible to compare 2 cohorts of patients in order to objectivize the contribution of manipulators to patient care, as the difficulty and time required to interpret RECIST 1.1 vary greatly from one patient to another, and depend mainly on the type of disease and its extent on the scanner.

Thus, 2 groups of patients comparable in terms of difficulty and interpretation time cannot be composed. For this reason, the study is based on the radiologist's assessment of the assistance provided by the MEM.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 and over
* Patient included in a clinical research protocol in oncology for solid cancer including RECIST 1.1 interpretation
* Disease measurable according to RECIST 1.1
* Patient not objecting to study participation
* Member of a social security scheme, or beneficiary of such a scheme.

Non inclusion Criteria:

* Patients with lymphoma or leukemia
* Patient contraindicated to iodinated contrast media injection
* Person in an emergency situation, adult subject to a legal protection measure (major under guardianship, curatorship or safeguard of justice), or unable to express, his/her non-opposition to participate in the study
* Unable to undergo medical follow-up for geographical, social or psychological reasons.

or psychological reasons.

Exclusion Criteria:

* Patient with renal insufficiency or allergy during the trial no longer allowing injection of iodinated contrast medium
* Patient refusing iodinated PDC injection during the study
* Patient withdrawn from the study including scanner interpretation in Recist 1.1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: major solid-cancer patient with baseline scan according to recists 1.1
Sampling Method: Probability Sample
Enrollment: 87 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Evaluate the pre-filling work on target and non-target lesions and the detection of any new lesions reported by the MEM trained in protocol evaluations in a structured table in order to prepare the radiologist's work in interpreting RECIST 1.1 scans. | up to 24 weeks
  Measurement of the rate of validation by the radiologist of the MEM's RECIST1.1 pre-analysis work, covering respectively assessment of target lesions, assessment of non-target lesions, detection of new lesions lesions, detection of new lesions and overall disease assessment on the first evaluation.

SECONDARY OUTCOMES:
Evaluate the benefit to the radiologist | up to 24 weeks
  Analysis of responses to radiologist questionnaires through a satisfaction survey created by our interdisciplinary team in economic and social sciences. There is no sharing of a common unit of measure, there is a only one questionnaire
Measure the MEM's expertise in identifying possible errors in the application of RECIST criteria to the Baseline review. | up to 24 weeks
  Measurement of the validation rate by the radiologist of the RECIST 1.1 retrospective critical analysis of the MEM of the Baseline examination.
Evaluate the benefit to the MEM | up to 24 weeks
  Analysis of responses to questionnaires completed by the MEM through a satisfaction survey created by our interdisciplinary team in economic and social sciences . There is no sharing of a common unit of measure, there is a only one questionnaire
Evaluate the benefits to the clinical research associate | up to 24 weeks
  Analysis of responses to questionnaires completed by the clinical research associate through a satisfaction survey created by our interdisciplinary team in economic and social sciences. There is no sharing of a common unit of measure, there is a only one questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Institut PAoli Camettes, Marseille, Institut Paoli Calmettes, France